CLINICAL TRIAL: NCT03196440
Title: Thresholds Analysis of Five Basic Tastes in the Elderly Population
Brief Title: Sensitivity of Basic Taste in Elderly
Acronym: TASTE
Status: Completed | Type: Observational
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49306815.0.0000.0071
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2016-07

CONDITIONS: Taste Disorders
Keywords: elderly; taste; thresholds
MeSH Terms: conditions — Taste Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to identify the thresholds sensitivity of the five basic tastes in an elderly population and relate to food intake, nutritional status, age, gender and others variables.

DETAILED DESCRIPTION:
The investigators propose a study of 300 elderly patients to characterize de sensitivity of the four basic tastes, according to the methodology of International Organization for Standardization (1985) and to identify umami taste (Mojet et al. 2001, 2003). This is a cross-sectional study. The length of the inclusion of the study will be 24 months. This study's general objective is: to characterize food intake, nutritional status and identify thresholds for the five basic tastes in an elderly population.

ELIGIBILITY:
Inclusion Criteria:

* 60 years old patient or older, who present oral feeding and the ability to express themselves to perform the sensory analysis tests will be included.

Exclusion Criteria:

* Patient with fever, flu, cold or some complication in the oral cavity will be excluded, since these factors can interfere in the perception of the tastes and those that do not present conditions to express themselves or deficits of cognition, being excluded the elderly that present result of the application of the Mini Mental under 24. In addition to those who do not agree to sign the Term of Free and Informed Consent.

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Threshold sensitivity is applied to determine the threshold of 5 basic tastes in elderly in ambulatory care. It is applied mini mental test to evaluate cognition, considering that those who presented a score equal to or greater than 24 points. A 24-hour recall was applied to check food intake. The mini nutritional assessment was applied to verify nutritional status. Other information, such as diagnoses and medications, were obtained from medical records. Information on socioeconomic parameters were obtained through a questionnaire applied to the patient.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2015-07-07 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

PRIMARY OUTCOMES:
Characterization of eldery according to sensitivity to basic tastes second age group and nutritional status | 3 years
  To identify the thresholds for detecting basic tastes in an elderly population and to relate to the age range and nutritional status.

CONTACTS AND LOCATIONS:
Overall Officials: Ilana E. Grinberg, PhD, Principal Investigator — Hospital Israelita Albert Einstein; Luciana DN Matos, PhD, Study Chair — Hospital Israelita Albert Einstein; Fabio GM Franco, PhD, Study Director — Hospital Israelita Albert Einstein
Locations (1):
- Ilana Elman Grinberg, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] ELMAN, I.; GERALDO, A. P. G. ; KARCHER, C. ; SILVA, Maria Elisabeth Machado Pinto e . Caracterização dos limiares de detecção do gosto umami em crianças com e sem câncer. Revista Brasileira de Crescimento e Desenvolvimento Humano, v. 23, p. 136, 2013.
- [Background] ELMAN, I.; SOARES, N. S. ; SILVA, Maria Elisabeth Machado Pinto e . Análise da Sensibilidade do Gosto Umami em Crianças com Câncer. Revista Brasileira de Cancerologia, v. 56, p. 237-242, 2010
- [Background] ELMAN, I.; SILVA, Maria Elisabeth Machado Pinto e . Crianças portadoras de Leucemia Linfóide Aguda: análise dos limiares de detecção dos gostos básicos segundo sexo. Revista Brasileira de Cancerologia, v. 53, p. 297-303, 2007.
- [Background] ELMAN, I.; SILVA, Maria Elisabeth Machado Pinto e . Crianças portadoras de câncer: sensibilidade ao PROP. Nutrição em Pauta, São Paulo, v. 4, n.79, p. 19-23, 2006.
- [Background] ELMAN, I.. Apoyo nutricional a los ninos con cáncer. Proyecto Felicidade, Washington, p. 43-45, 2006.
- [Background] SILVA, Maria Elisabeth Machado Pinto e ; PATON, Ive ; TRIGO, Marlene ; ELMAN, I. . Perfis socioeconômico e nutricional de crianças e adolescentes com câncer. Revista Brasileira de Nutrição Clínica, São Paulo, v. 19, n.3, p. 123-127, 2004.
- [Background] GALDOLFO, Adriana S ; VIEIRA, Maria Aparecida ; ELMAN, I. . Oncologia. In: Ana Paula Alves da Silva; GA Corradi; Patricia Zamberlam. (Org.). Manual de dietas hospitalares em pediatria: Guia de Conduta Nutricional
- [Background] Elman I. Cancer bearer children: Thresholds analysis of basic taste detection and sensivity to 6-n-propylthiouracil. São Paulo; 2005. [Dissertação de Mestrado - Faculdade de Saúde Pública da USP].
- [Background] Elman I. Characterization of childen with câncer according to sensivity to umami and food consumption. [Tese de Doutorado em Nutrição e Saúde Pública]. São Paulo: Faculdade de Saúde Pública da USP; 2011.
- [Result] Grinberg IE, de Mello Franco FG, Machado Pinto-e-Silva ME, Janot Matos LDN. Are there relationships between basic tastes, age, gender and nutritional status in an elderly population? World Journal of Advanced Research and Reviews, 2020, 07(02), 285-293
- See also: Lattes — http://lattes.cnpq.br/6963575752679160